CLINICAL TRIAL: NCT04304482
Title: ANAVEX2-73-RS-003 is a Phase 2/3, Double-blind, Randomized, Placebo-controlled Safety and Efficacy Study in Pediatric Patients With RTT
Brief Title: ANAVEX2-73 Study in Pediatric Patients With Rett Syndrome
Acronym: EXCELLENCE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: Anavex Australia Pty Ltd. (Industry); Anavex Germany GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX2-73-RS-003
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ANAVEX2-73 Active (Experimental): ANAVEX2-73 liquid oral solution
  Interventions: Drug: ANAVEX2-73 oral liquid
- ANAVEX2-73 Placebo (Placebo Comparator): Placebo liquid oral solution
  Interventions: Drug: Placebo oral liquid

INTERVENTIONS:
Drug: ANAVEX2-73 oral liquid — Liquid oral solution
  Other Names: Blarcamesine
  Arms: ANAVEX2-73 Active
Drug: Placebo oral liquid — Liquid oral solution
  Arms: ANAVEX2-73 Placebo

SUMMARY:
ANAVEX2-73-RS-003 is a Phase 2/3, double-blind, randomized, placebo-controlled dose escalation safety, tolerability and efficacy study in patients 5-17 years of age with RTT using endpoints including multiple clinical and exploratory molecular and biochemical measures.

DETAILED DESCRIPTION:
This Phase 2/3 efficacy study is designed as a double-blind, randomized, placebo-controlled study.

This is a 12-week placebo-controlled study of ANAVEX2-73 oral solution for the treatment of patients with RTT 5-17 years of age. A voluntary option will be offered for all patients who meet the exposure criteria for ANAVEX2-73 to continue a 48-week open label extension.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 5 years to 17 (inclusive).
* Diagnosis of classic RTT, according to 2010 criteria, and a MECP2 mutation.
* Post-regression stage, defined as ≥ 6 months since last loss of spoken language or motor (fine or gross) skills.
* Clinical Global Impression - Severity (CGI-S) score of 4 or greater at Screening.
* Current pharmacological treatment regimen, including supplements, has been stable for at least 4 weeks.
* If on AEDs, 1-4 AEDs allowed. Treatment must be stable (drug, dose, interval of administration) for 30 days prior to enrollment.
* If the subject is already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, participation in these programs must have been continuous during the 90 days prior to the screening visit and subjects or their parent/caregiver/LAR will not electively initiate new or modify ongoing interventions for the duration of the study.
* The subject's caregiver/LAR is English-speaking and has sufficient language skills to complete the caregiver assessments and has the ability to keep accurate seizure diaries.
* If participant is a woman of childbearing potential (WOCBP#), a negative urine or serum pregnancy test is required to confirm she is not pregnant.
* Prior to the conduct of study-specific procedures, the subject's parent/caregiver/LAR must provide written informed consent. If applicable, the research team must attempt to obtain consent from both parents.

Exclusion Criteria:

* Patients who have a progressive medical or neurological condition that in the opinion of the Investigator would interfere with the conduct of the study.
* Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
* History or clinically evident neurologic (e.g., head trauma with loss of consciousness) or psychiatric condition that the Investigator deems may interfere with interpretability of data.
* Indication of liver disease, defined by serum levels of ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3x upper limit of normal (ULN) as determined during screening.
* Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years.
* Other clinically significant abnormality on physical, neurological, laboratory, or electrocardiogram (ECG) examination (e.g., long QT) that could compromise the study or be detrimental to the participant.
* Any known hypersensitivity to any of the excipients contained in the study drug or placebo formulation.
* Other co-morbid or chronic illness beyond that known to be associated with RTT.
* Subjects who plan to initiate or change pharmacologic or nonpharmacologic intervention during the course of the study.
* Subjects taking another investigational drug currently or within the last 30 days.
* Any other criteria (such as a clinically significant screening blood test result), which in the opinion of the Investigator could interfere with the study conduct or outcome.
* Treatment with strong inhibitors or inducers of CYP3A4 or CYP2C19 is not stable (drug, dose) for 30 days prior to screening. Although these medications are not excluded, caution is advised when enrolling participants on potent CYP3A4 or CYP2C19 inducers or inhibitors (see respective section).
* Patients with hepatic and renal impairment.

Ages: 5 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
RSBQ | 12 weeks
  Change from baseline to End of Treatment (EOT) in the Rett Syndrome Behaviour Questionnaire (RSBQ) Total score
Incidents of Adverse Events | 12 weeks
  Change from baseline to End of Treatment (EOT)

SECONDARY OUTCOMES:
CGI-I | 12 weeks
  Change from baseline to End of Treatment (EOT) in the Clinical Global Impression Improvement Scale (CGI-I) score
Anxiety, Depression, and Mood Scale (ADAMS) | 12 weeks
  Anxiety, Depression, and Mood Scale (ADAMS)
Motor Behavioral Assessment-7 dynamic pediatric items (MBA-Ped7) | 12 weeks
  Motor Behavioral Assessment-7 dynamic pediatric items (MBA-Ped7)
Children's Sleep Habits Questionnaire (CSHQ) | 12 weeks
  Children's Sleep Habits Questionnaire (CSHQ)
Seizure Frequency via seizure diary | 12 weeks
  Seizure Frequency via seizure diary
Incidence of Adverse Events | 12 weeks
  Incidence of Adverse Events
RSBQ Emotional Factor-Pediatric (subset of the RSBQ) | 12 weeks
  RSBQ Emotional Factor-Pediatric (subset of the RSBQ)
Rett Syndrome Caregiver Inventory Assessment (RTT CIA) | 12 weeks
  Rett Syndrome Caregiver Inventory Assessment (RTT CIA)
Child Health Questionnaire-Parent Form 50 (CHQ-PF50) | 12 weeks
  Child Health Questionnaire-Parent Form 50 (CHQ-PF50)

OTHER OUTCOMES:
Glutamate Plasma Concentration | 12 weeks
  Glutamate Plasma Concentration
GABA Plasma Concentration | 12 weeks
  GABA Plasma Concentration
Genetic variant SIGMAR1, COMT | 12 weeks
  Genetic variant SIGMAR1, COMT
Maximum Plasma Concentration [Cmax] | 12 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Maximum Plasma Concentration [Cmax] relationship with RSBQ | 12 weeks
  Number of participants with positive Maximum Plasma Concentration [Cmax] relationship with RSBQ
Other Amino Acid Plasma concentrations | 12 weeks
  Other Amino Acid Plasma concentrations
Measure of gene DNA variants and gene RNA expressions | 12 weeks
  Number of participants with active dose compared gene DNA variants and gene RNA expressions

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (3):
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Austin Health, Melbourne, Victoria
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital LHSC, London, Ontario
  - Holland Bloorview Kids Hospital, Toronto, Ontario
- United Kingdom (5):
  - Royal Hospital for Children, Edinburgh
  - Evelina London Children's Hospital, London
  - King's College of London, London
  - Manchester CGM, St Mary's Hospital, Manchester
  - Nottingham University Hospital NHS Trust, Nottingham

REFERENCES:
- [Derived] Heussler HS. Emerging Therapies and challenges for individuals with Angelman syndrome. Curr Opin Psychiatry. 2021 Mar 1;34(2):123-128. doi: 10.1097/YCO.0000000000000674. PMID 33395098